CLINICAL TRIAL: NCT02137694
Title: Comparison of the Urinary and Vaginal Auto-takings for the Research for Papillomavirus as the Examination of Orientation in the Organized Screening of the Cervical Cancer.
Brief Title: Research for Papillomavirus as the Examination of Orientation in the Organized Screening of the Cervical Cancer
Acronym: PapU-APV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RB 13.161 PapU-APV
Record Dates: First submitted 2014-04-30; First posted 2014-05-14 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2015-12

CONDITIONS: Research Human Papillomavirus ( HPV) by Vaginal Auto-takings ( APV) and Urinary Test
Keywords: Papillomavirus; Vaginal auto-takings; Urinary test
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PapU-APV (Other): No drug and no placebo will be used in this study. For the study participants, only their medical history data and vaginal auto-takings ( APV) and urinary will be collected.
  Interventions: Other: vaginal auto-takings and urinary test

INTERVENTIONS:
Other: vaginal auto-takings and urinary test — vaginal auto-takings and urinary test

SUMMARY:
Auto-takings by APU and vaginal APV during the consultations for FCU in the department of gynecology-obstetrics (Group 1) according to an instructions for use proposed to the inclusive women, with consent; the same proposal, APU and APV, is made for other consultations requiring a screening on the CHRU (Group 2: dermatology, endocrinology, ambulatory surgery, inner medicine, pneumology, oncology). Auto-takings transmitted in the laboratory of the CHRU of Brest for test HPV by quantitative real-time PCR. Results transmitted to the women and to the doctors of consultation. In case of positive test (15 %), the patients are directed to a gynecologist. Confrontation with the cytological data when available (Group 1) .

ELIGIBILITY:
Inclusion Criteria:

* All the 25-65-year-old women requiring a screening and seen in consultation of the departments targeted by the CHRU of Brest

Exclusion Criteria:

* Women except age limit, refusal to participate, hysterectomy, pregnancy and post-therapeutic follow-up.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Research for human Papillomavirus by vaginal auto-takings and urinary test | 6 months
  Estimate the research for human Papillomavirus ( HPV) in the vaginal auto-takings ( APV) and urinary ( APU) test at women from 25 to 65 years old requiring a screening.

SECONDARY OUTCOMES:
The global logistic of the study | 6 months
  Estimate the practicability, the organization of the screening, the follow-up of the women at the Brest Hospital and at Landerneau Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Christopher PAYAN, PU-PH, Principal Investigator — CHRU Brest
Locations (2):
- France (2):
  - CHRU de Brest, Brest, France
  - Hôpital Ferdinand Grall, Landerneau, France